CLINICAL TRIAL: NCT02040103
Title: Prophylaxis of Thromboembolism in Critically Ill Patients Using Combined Intermittent Pneumatic Compression(IPC) and Pharmacologic Prophylaxis Versus Pharmacologic Prophylaxis Alone: A Multicenter Randomized Controlled Trial
Brief Title: Pneumatic Compression for Preventing Venous Thromboembolism
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: King Abdulaziz Medical City, Jeddah (Unknown); King Abdulaziz Hospital, Al Ahsa (Unknown); Unity Health Toronto (Other); King Fahad Medical City (Other Government); Assir Central Hospital (Unknown); Royal North Shore Hospital (Other); Mount Sinai Hospital, Canada (Other); Prince Sultan Military Medical City (Other); King Faisal Specialist Hospital & Research Center (Other); Gosford Hospital, Australia (Unknown); St Vincent's Hospital - Sydney, Australia (Other); Medanta, The Medicity, India (Other); King Fahad Hospital of the University, Al Khobar (Unknown); King George's Medical University, India (Unknown)
Responsible Party: Principal Investigator, Dr Yaseen Arabi, Chairman, Intensive Care Department, King Abdulaziz Medical City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC12-045
Record Dates: First submitted 2013-11-03; First posted 2014-01-20 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep Vein Thrombosis; Pulmonary Embolism; Intermittent Pneumatic Compression; Pharmacologic DVT; Prophylaxis; Critically Ill Patients.
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Pneumatic Compression(IPC) (Experimental): The intervention group will be receiving Intermittent Pneumatic Compression(IPC)
  Interventions: Device: pneumatic compression
- No Intermittent Pneumatic Compression (No Intervention): patients will not receive Intermittent Pneumatic Compression

INTERVENTIONS:
Device: pneumatic compression — All IPC devices intended for DVT prophylaxis are acceptable in the study. Sequential devices (cuffs have several chambers) are preferred, but non-sequential (cuffs have single chambers) are acceptable.
  Arms: Intermittent Pneumatic Compression(IPC)

SUMMARY:
Patients admitted to the intensive care unit are at high risk of developing clots in the veins of the lower extremities. The objective of this study is to examine whether the use of a device that provides intermittent compression to the legs in addition to the use of low-dose blood thinners, provides an additional protection when compared to the use of blood thinners alone. Patients who are admitted to the intensive care unit are receiving low-dose blood thinners to prevent clots are candidates for this study. Patients who are enrolled will continue to receive blood thinners but some will additionally receive the leg compression. The additional use of leg compression may provide protection from clots. The main side effect is possible skin abrasions but this is usually mild. The study is sponsored by King Abdullah International Medical Research Center(KAIMRC) and King Abdulaziz City for Science and Technology(KACST) and will be conducted in several hospitals in Saudi Arabia, Canada, Australia, Brazil and possibly other countries. The study started July 2014 and is to continue for 4 years.

DETAILED DESCRIPTION:
There is no randomized controlled trial examining effect of the adjunct use of IPC with pharmacologic prophylaxis compared to pharmacologic prophylaxis (UFH, LMWH) alone in critically ill patients for VTE prevention.

ELIGIBILITY:
INCLUSION CRITERIA

A. Medical-Surgical ICU patients >14 years old at participating ICU. ICUs that use other age cut-off for adult patients will adhere to their local standard (16 or 18 years) B. Weight > 45kg C. Expected ICU LOS> 72hrs D. Eligible for pharmacologic thromboprophylaxis with UFH and LMWH.

EXCLUSION CRITERIA

A. Patient treated with IPC for > 24 hours in this current ICU admission. B. Patient in the ICU> 48 hours. C. Patient treated with pharmacologic VTE prophylaxis with medications other than UFH or LMWH.

D. Inability or contraindication to applying IPC to both legs i.Burns in the lower extremities, lacerations, active skin infection, & ischemic limb in the legs at the site of IPC placement ii. Acute ischemia in the lower extremities iii. Amputated foot or leg on one or two sides iv. Compartment Syndrome v. Severe peripheral arterial disease vi. Vein ligation, gangrene, recent vein grafts, and draining incisions vii. Evidence of bone fracture in lower extremities E. Therapeutic dose of anticoagulation with UFH or LMWH F. Pregnancy G. Limitation of life support, life expectancy < 7 days or palliative care H. Allergy to the sleeves material I. Patients with Inferior Vena Cava (IVC) Filter

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Proximal deep vein thrombosis(DVT) diagnosed by compression ultrasound | 28 days from randomization
  The primary outcome is incident proximal leg DVT, defined as detected 3 or more days post-randomization and up to ICU discharge or day 28 post randomization

SECONDARY OUTCOMES:
Pulmonary Embolism | from the time of randomization to 90 days
  Pulmonary Embolism: will be followed up to ICU discharge or day 28 post randomization.
  ICU Mortality. Death in ICU during the same ICU admission. Hospital Mortality. Death in the hospital (in ICU or on ward) during the same hospital admission. (Hospital mortality will be censored at 1 year from the date of enrollment).
  28-day Mortality: Death before or at day 28 of enrollment. 90-day Mortality: Death before or at day 90 of enrollment.

OTHER OUTCOMES:
ICU Length of stay and duration of mechanical ventilation | Number of days in ICU with an average expected duration of 10 days and number of days of mechanical ventillation with an expected average duration of 8 days.
  ICU Length of stay: Number of calendar days between admission and discharge from ICU.
  Duration of mechanical ventilation: Number of calendar days between start and end of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen Arabi, MD, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- Intensive Care Unit, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Al-Dorzi HM, Arishi H, Al-Hameed FM, Burns KEA, Mehta S, Jose J, Alsolamy SJ, Abdukahil SAI, Afesh LY, Alshahrani MS, Mandourah Y, Almekhlafi GA, Almaani M, Al Bshabshe A, Finfer S, Arshad Z, Khalid I, Mehta Y, Gaur A, Hawa H, Buscher H, Lababidi H, Al Aithan A, Al-Dawood A, Arabi YM; Saudi Critical Care Trials Group. Performance of Risk Assessment Models for VTE in Patients Who Are Critically Ill Receiving Pharmacologic Thromboprophylaxis: A Post Hoc Analysis of the Pneumatic Compression for Preventing VTE Trial. Chest. 2025 Feb;167(2):598-610. doi: 10.1016/j.chest.2024.07.182. Epub 2024 Sep 2. PMID 39232999
- [Derived] Al-Dorzi HM, AlQahtani S, Al-Dawood A, Al-Hameed FM, Burns KEA, Mehta S, Jose J, Alsolamy SJ, Abdukahil SAI, Afesh LY, Alshahrani MS, Mandourah Y, Almekhlafi GA, Almaani M, Al Bshabshe A, Finfer S, Arshad Z, Khalid I, Mehta Y, Gaur A, Hawa H, Buscher H, Lababidi H, Al Aithan A, Arabi YM; Saudi Critical Care Trials Group. Association of early mobility with the incidence of deep-vein thrombosis and mortality among critically ill patients: a post hoc analysis of PREVENT trial. Crit Care. 2023 Mar 3;27(1):83. doi: 10.1186/s13054-023-04333-9. PMID 36869382
- [Derived] Al-Dorzi HM, Al-Dawood A, Al-Hameed FM, Burns KEA, Mehta S, Jose J, Alsolamy S, Abdukahil SAI, Afesh LY, Alshahrani MS, Mandourah Y, Almekhlafi GA, Almaani M, Al Bshabshe A, Finfer S, Arshad Z, Khalid I, Mehta Y, Gaur A, Hawa H, Buscher H, Lababidi H, Al Aithan A, Arabi YM. The effect of intermittent pneumatic compression on deep-vein thrombosis and ventilation-free days in critically ill patients with heart failure. Sci Rep. 2022 May 20;12(1):8519. doi: 10.1038/s41598-022-12336-9. PMID 35595804
- [Derived] Arabi YM, Burns KEA, Alsolamy SJ, Alshahrani MS, Al-Hameed FM, Arshad Z, Almaani M, Hawa H, Mandourah Y, Almekhlafi GA, Al Aithan A, Khalid I, Rifai J, Rasool G, Abdukahil SAI, Jose J, Afesh LY, Al-Dawood A; Saudi Critical Care Trials Group. Surveillance or no surveillance ultrasonography for deep vein thrombosis and outcomes of critically ill patients: a pre-planned sub-study of the PREVENT trial. Intensive Care Med. 2020 Apr;46(4):737-746. doi: 10.1007/s00134-019-05899-1. Epub 2020 Feb 24. PMID 32095845
- [Derived] Arabi YM, Al-Hameed F, Burns KEA, Mehta S, Alsolamy SJ, Alshahrani MS, Mandourah Y, Almekhlafi GA, Almaani M, Al Bshabshe A, Finfer S, Arshad Z, Khalid I, Mehta Y, Gaur A, Hawa H, Buscher H, Lababidi H, Al Aithan A, Abdukahil SAI, Jose J, Afesh LY, Al-Dawood A; Saudi Critical Care Trials Group. Adjunctive Intermittent Pneumatic Compression for Venous Thromboprophylaxis. N Engl J Med. 2019 Apr 4;380(14):1305-1315. doi: 10.1056/NEJMoa1816150. Epub 2019 Feb 18. PMID 30779530
- [Derived] Arabi Y, Al-Hameed F, Burns KEA, Mehta S, Alsolamy S, Almaani M, Mandourah Y, Almekhlafi GA, Al Bshabshe A, Finfer S, Alshahrani M, Khalid I, Mehta Y, Gaur A, Hawa H, Buscher H, Arshad Z, Lababidi H, Al Aithan A, Jose J, Abdukahil SAI, Afesh LY, Dbsawy M, Al-Dawood A; PREVENT trial Group. Statistical analysis plan for the Pneumatic CompREssion for PreVENting Venous Thromboembolism (PREVENT) trial: a study protocol for a randomized controlled trial. Trials. 2018 Mar 15;19(1):182. doi: 10.1186/s13063-018-2534-6. PMID 29544550
- [Derived] Arabi YM, Alsolamy S, Al-Dawood A, Al-Omari A, Al-Hameed F, Burns KE, Almaani M, Lababidi H, Al Bshabshe A, Mehta S, Al-Aithan AM, Mandourah Y, Almekhlafi G, Finfer S, Abdukahil SA, Afesh LY, Dbsawy M, Sadat M. Thromboprophylaxis using combined intermittent pneumatic compression and pharmacologic prophylaxis versus pharmacologic prophylaxis alone in critically ill patients: study protocol for a randomized controlled trial. Trials. 2016 Aug 3;17(1):390. doi: 10.1186/s13063-016-1520-0. PMID 27488380